CLINICAL TRIAL: NCT05991388
Title: A Global Study of Novel Agents in Paediatric and Adolescent Relapsed and Refractory B-cell Non-Hodgkin Lymphoma
Acronym: Glo-BNHL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Cancer Research UK (Other); Fight Kids Cancer (Other); Regeneron Pharmaceuticals (Industry); ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_21-124; ITCC-100 (Other: ITCC); 1004701 (Other: IRAS ID)
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — loncastuximab tesirine; Rituximab; Ifosfamide; Carboplatin; Etoposide; etoposide phosphate; Dexamethasone; Immunotherapy, Adoptive; Tubercidin

STUDY DESIGN:
Intervention Model Description: Platform trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment Arm I - BsAb - Odronextamab (Experimental): Patients will receive odronextamab given as an intravenous infusion weekly for 12 weeks, then every two weeks until nine months, and every four weeks thereafter until progression or for a maximum of two years
  Interventions: Drug: Odronextamab
- Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE (Experimental): Patients will receive loncastuximab tesirine given as a 30-minute intravenous infusion with each cycle of modified R-ICE (maximum three cycles)
  Interventions: Drug: Loncastuximab tesirine; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Etoposide Phosphate; Drug: Dexamethasone
- Treatment Arm III - CAR T-cells - TBC (Experimental): Patients will receive CAR-T cell therapy - agent TBC
  Interventions: Biological: CAR T-cells (TBC)

INTERVENTIONS:
Drug: Odronextamab — CD20xCD3 bispecific antibody
  Other Names: REGN-1979
  Arms: Treatment Arm I - BsAb - Odronextamab
Drug: Loncastuximab tesirine — CD-19-directed antibody-drug conjugate
  Other Names: ADCT-402
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Drug: Rituximab — Modified R-ICE chemotherapy
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Drug: Ifosfamide — Modified R-ICE chemotherapy
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Drug: Carboplatin — Modified R-ICE chemotherapy
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Drug: Etoposide — Modified R-ICE chemotherapy
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Drug: Etoposide Phosphate — Modified R-ICE (Treatment Arm II)
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Drug: Dexamethasone — Modified R-ICE chemotherapy
  Arms: Treatment Arm II - ADC with Standard Chemotherapy - Loncastuximab tesirine with modified R-ICE
Biological: CAR T-cells (TBC) — Modified R-ICE chemotherapy
  Arms: Treatment Arm III - CAR T-cells - TBC

SUMMARY:
The Glo-BNHL trial is trying to find better medicines for children and young people with B-cell non-Hodgkin Lymphoma (B-NHL) that does not go away (refractory B-NHL) or does but comes back again (relapsed B-NHL). B-NHL is a type of cancer that develops inside or outside of lymph nodes (glands) and organs such as the liver or spleen. Examples of B-NHL are Burkitt Lymphoma and Diffuse Large B Cell Lymphoma, which may be other names used to describe this type of cancer. It is very difficult to cure relapsed or refractory B-NHL. The medicines used now are very powerful with many side effects and only cure around 30 in every 100 children treated. It is very important that investigators quickly find better medicines for these children and young people.

The Glo-BNHL trial will include three groups of children and young people, each given a new medicine (either alone or with chemotherapy). The investigators are looking to make sure the new medicines are safe and that they work to treat the cancer. If the medicine in one group does not work for a child in the trial, then they may be able to join a different group to have another new medicine.

Experts from around the world will carefully pick the medicines most likely to be helpful to be part of the trial. If one of the new medicines seems not to be working as well as hoped then the investigators will take it out of the trial as soon as possible. This will let other new medicines be added to the trial and tested. If a medicine does seem to be working well, then it will continue in the trial to make sure it really is the most useful medicine available.

Children from around the world will be invited to take part in the trial. The investigators will then check on them for at least two years after they finish the trial treatment to look for possible side effects of the new medicine.

DETAILED DESCRIPTION:
Glo-BNHL is an adaptive prospective international multicentre platform clinical trial designed to evaluate the safety and efficacy of novel agents for the treatment of children, adolescents, and young adults with relapsed and/or refractory B-cell non-Hodgkin Lymphoma (r/r BNHL). The trial is designed to generate sufficient evidence to potentially be practice-changing in this rare cancer setting. With the trial incorporating an initial stage evaluating efficacy followed potentially by an expansion stage to provide confirmatory analysis, the trial could be considered to be phase II/III.

Novel agents will be prioritised for inclusion in the platform according to an overarching prioritisation list and a robust systematic scientific assessment, performed by the international Trial Steering Committee (TSC).

The platform consists of three parallel treatment arms, each one investigating a different novel agent in a group of patients. The platform allows the testing of a pipeline of novel agents in each treatment arm consecutively. Patients in the platform may be enrolled into any of the available treatment arms for which they are eligible. The classes of novel agents prioritised for inclusion at the initiation of the trial are:

* Treatment Arm I: Bispecific antibodies (BsAbs)
* Treatment Arm II: Antibody-drug conjugates (ADC) with standard chemotherapy
* Treatment Arm III: Chimeric antigen receptor (CAR) T-cells

The platform trial has an adaptive Bayesian design that facilitates efficient GO/NoGO decisions relevant to the target population enrolled in each treatment arm. The Bayesian approach estimates the probability that a novel agent is clinically effective and enables decision-making even with small numbers of patients. It can also incorporate prior knowledge, thereby maximising the utility of all available data in this rare population. It facilitates continuous evaluation of any novel agent as the sample size increases.

Furthermore it allows for the discontinuation of an agent if the observed trial data demonstrate a high probability that the novel agent is ineffective at any time, allowing the next agent in the pipeline to be introduced. If the prioritisation of classes of novel agents by the TSC changes, treatment arms can be amended, added, or removed to reflect this. Not all Treatment Arms will necessarily be open to recruitment at all times.

ELIGIBILITY:
Inclusion criteria applicable to all treatment arms:

* Histologically proven mature B-NHL (Diffuse Large B-Cell Lymphoma (DLBCL), Burkitt Lymphoma/Leukaemia or atypical Burkitt/Burkitt-like lymphoma, primary mediastinal large B-cell lymphoma (PMLBL), and mature B-NHL/Not Otherwise Specified (NOS)) at initial diagnosis
* Radiologically and/or histologically proven B-NHL in first relapse (only one prior line of therapy) or subsequent relapse (more than one prior line of therapy) or refractory(*) B-NHL. (Note: relapses following prior targeted therapy must have continuing target positivity, confirmed by an established method).
* If relapse occurs more than two years after previous therapy, a biopsy must be performed
* Evaluable disease as per the international paediatric non-Hodgkin Lymphoma response criteria, including:

  * at least one bi-dimensionally measurable nodal lesion >1.5 cm in its longest dimension;
  * or at least one bi-dimensionally measurable extra-nodal lesion >1.0 cm in its longest dimension on computerised tomography (CT) or Magnetic Resonance Imaging (MRI);
  * or bone marrow involvement (≥25% involvement from bone marrow, if only site of disease. Any standard method of assessment is acceptable i.e. cytomorphology, flow cytometry and/or immunohistochemistry);
  * or, dependent on treatment arm, evaluable Central Nervous System (CNS) only disease (evaluable by imaging or Cerebrospinal Fluid (CSF) analysis)(**)
* Age from birth to ≤25 years old at the time of trial entry
* Performance status ≥50 using Karnofsky or Lansky performance scores
* Life expectancy of ≥8 weeks
* Adequate bone marrow function documented by:

  * Platelet count ≥50x 10^9/L (no platelet transfusion therapy within seven days prior to treatment) unless bone marrow involvement(***)
  * Absolute neutrophil count (ANC) ≥0.75 x 10^9/L (no granulocyte colony stimulating factor within 2 days prior to treatment) unless bone marrow involvement(***)
* Adequate hepatic function documented by:

  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤5 x upper limit of normal (ULN)
  * Total bilirubin ≤1.5 X ULN ***Patients with known Gilbert syndrome will be excluded if the total bilirubin value is >4 x ULN for the local general population
* Documented negative pregnancy test for female patients of childbearing potential within seven days prior to trial entry
* Patients of reproductive potential agrees to use effective contraception whilst on trial treatment and for 12 months following treatment discontinuation
* Written informed consent given by patient and/or parents/legal representative

Inclusion criteria applicable to treatment arm I only:

* Male patients of reproductive potential must agree not to donate sperm whilst on trial treatment and for 6 months following treatment discontinuation
* Adequate renal function, creatinine clearance >45 ml/min by measurement or estimation (if creatinine levels are normal for the patient's age, using the Cockroft-Gault Equation is sufficient)
* For patients with bone marrow involvement(***) or splenic sequestration, adequate bone marrow function documented by:

  * Platelet count ≥25 x 10^9/L (no platelet transfusion therapy within three days prior to treatment)
  * Haemoglobin level ≥7 g/dL
  * Absolute neutrophil count (ANC) ≥0.5 x 10^9/L (no granulocyte colony stimulating factor within two days prior to treatment)
* Patients who have received CAR T-cell therapy or other cellular therapies more than 28 days prior must demonstrate recovery from acute toxicities and have measurable disease

Inclusion criteria applicable to treatment arm II only:

* Adequate renal function, by measured glomerular filtration rate (GFR) >60 ml/min/1.73m^2 (estimated GFR is not sufficient)
* For patients with bone marrow involvement(***) or splenic sequestration, requirements for bone marrow function do not apply

(*) Refractory disease

The following patients are considered to have refractory disease and can be included in this trial:

* Patients with who do not achieve PR or CR with last therapy
* Patients with partial response to last therapy (biopsy proven), with no evidence of progression

(**) CNS only disease Patients with CNS only disease may be eligible depending on the treatment arm. Please refer to the relevant treatment arm specific eligibility criteria.

(***) Bone marrow involvement Patients who have ≥ 25% blasts in the bone marrow are considered to have bone marrow involvement. For these patients, requirements for bone marrow function are dependent on treatment arm. Please refer to the relevant treatment arm specific eligibility criteria.

Exclusion Criteria:

* B-cell Acute Lymphoblastic Leukaemia (B-ALL)/B-cell Lymphoblastic Lymphoma (B-LBL)
* Patients within:

  * 90 days after an allogenic HSCT procedure
  * 45 days after an autologous HSCT procedure
  * 28 days of experiencing graft versus host disease (GvHD) requiring systemic therapy, and/or immunosuppressive treatment
  * 14 days of previous investigational treatment
  * 28 days of receiving craniospinal radiation; or 14 days of any other radiation
  * For patients who have received any CAR T-cell therapy or other cellular therapies, see treatment arm specific eligibility criteria
* Patients who have ongoing acute toxicities from most recent lymphoma directed therapy
* Patients with known DNA repair disorder or known primary immunodeficiency
* Patients who are pregnant or breastfeeding (exclusively or partially)
* Patients who cannot regularly be followed up in accordance with the protocol due to psychological, social, geographical or other issues
* Patients for whom non-compliance with treatment or trial procedures is expected
* Uncontrolled concomitant infection. Severe infection (such as sepsis, pneumonia, etc.) should be clinically controlled at the time of trial entry
* Known HIV positivity
* Hepatitis B carrier status, history of Hepatitis B Virus or positive serology. A patient is considered as a Hepatitis B Virus carrier or to have (had) Hepatitis B Virus infection in case of:

  * Unimmunized and HBsAg and/or anti-HBs antibody and/or anti- HBc antibody positive,
  * Immunized and HBsAg and/or anti-HBc antibody positive.
* Live vaccine within 28 days prior to trial entry
* Known history of hypersensitivity to any of the treatments or excipients

Exclusion criteria applicable to treatment arm I only:

* Central Nervous System (CNS) only disease
* Patients within 28 days of any CAR-T cell therapy or other cellular therapies
* Left ventricular shortening fraction (LVSF) <27% or left ventricular ejection fraction (LVEF) <50%, as determined by ECHO or MUGA, any evidence of pericardial effusion (except trace or physiological) as determined by an ECHO, and any clinically significant arrhythmias
* Known CD20 negative disease at initial diagnosis
* Seizure within the last 12 months
* Prior treatment with CD20 x CD3 bispecific therapy
* Known hypersensitivity to both allopurinol and rasburicase

Exclusion criteria applicable to treatment arm II only:

* Patients within 42 days of any CAR-T cell therapy or other cellular therapies
* Clinically significant (Grade ≥2) third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* Steroid treatment for more than a total of seven days in the 14 days prior to trial entry

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Arm I: BsAb: Occurrence of an objective response (OR) | At the end of week 12 of treatment
  Occurrence of an objective response (OR) i.e. Complete Response (CR) or Partial Response (PR) after 12 weeks of treatment assessed by Independent Central Review (according to International Paediatric Non-Hodgkin Lymphoma Response Criteria)
Treatment Arm II: ADC with standard chemotherapy: Occurrence of CR | At the end of Cycle 2 and Cycle 3 of treatment (each cycle is 28 days)
  Occurrence of CR within a maximum of three cycles of treatment assessed by Independent Central Review (according to International Paediatric Non-Hodgkin Lymphoma Response Criteria)

SECONDARY OUTCOMES:
Event-free survival time (EFS) | From start of treatment until last patient has been followed up for 2 years
  All treatment arms
Progression-free survival time (PFS) | From start of treatment until last patient has been followed up for 2 years
  All treatment arms
Overall survival time (OS) | From start of treatment until last patient has been followed up for 2 years
  All treatment arms
Best overall response (BOR) during treatment | At the end of weeks 4, 8, and 12 for Treatment Arm I; at the end of cycles 1, 2, and 3 for Treatment Arm II (each cycle is 28 days)
  All treatment arms
Duration of response (DOR) | From start of treatment until last patient has been followed up for 2 years
  All treatment arms
Occurrence of an objective response (OR), where relevant | At the end of cycles 1, 2, and 3 (each cycle is 28 days)
  Treatment arm specific
Occurrence of adverse events of special interest (AESI) | From start of treatment until 90 days after last day of treatment
  Treatment arm specific
Occurrence of treatment emergent adverse events (TEAEs), where relevant | From start of treatment until 90 days after last dose
  Treatment arm specific

CONTACTS AND LOCATIONS:
Overall Officials: Amos Burke, Principal Investigator — University of Birmingham
Locations (11):
- Australia (3):
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- St. Anna Children's Hospital, Vienna, Austria
- UZ Leuven, Leuven, Belgium
- Princess Máxima Centre for Pediatric Oncology, Utrecht, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No